CLINICAL TRIAL: NCT06785987
Title: Continuous Lidocaine Infusion in Thyroid Surgery Using Intraoperative Neurophysiological Monitoring
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Sun Huai-Jhih, Anesthesiologist, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KSVGH24-CT1-12 2024.2.7
Record Dates: First submitted 2025-01-10; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Thyroid Disease; Thyroid Surgery; Lidocaine Infusion
Keywords: lidocaine; Thyroid surgery
MeSH Terms: conditions — Thyroid Diseases | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant
Masking Description: The Participant will be under general anesthesia, masking the Participant from knowing the exact drugs using during the surgery.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- intermittent fentanyl infusion (Active Comparator): Maintained with volatile anesthetic gas (sevoflurane) and intermittent fentanyl infusion.
  Interventions: Drug: intermittent fentanyl infusion
- Continuous Lidocaine Infusion (Experimental): Maintained with sevoflurane and continuous lidocaine infusion under dosage: 1.5 mg/kg/hr
  Interventions: Drug: Continuous Lidocaine Infusion
- Continuous remifentanil Infusion (Active Comparator): Maintained with sevoflurane and continuous remifentanil infusion under dosage: 3-5μg /kg/hr
  Interventions: Drug: Continuous remifentanil Infusion

INTERVENTIONS:
Drug: Continuous Lidocaine Infusion — Maintained with sevoflurane and continuous lidocaine infusion under dosage: 1.5 mg/kg/hr
  Other Names: Lidocaine
  Arms: Continuous Lidocaine Infusion
Drug: intermittent fentanyl infusion — Maintained with volatile anesthetic gas (sevoflurane) and intermittent fentanyl infusion.
  Arms: intermittent fentanyl infusion
Drug: Continuous remifentanil Infusion — Maintained with sevoflurane and continuous remifentanil infusion under dosage: 3-5μg /kg/hr
  Arms: Continuous remifentanil Infusion

SUMMARY:
Thyroid surgery is a common procedure for the treatment of thyroid tumors, nodules and other related lesions. During this procedure, intraoperative neurophysiological monitoring is used to protect the recurrent laryngeal nerves. For the nerve monitor to work properly, a reduced muscle relaxant dosage is indicated. The main objectives of the anesthesiologist are maintaining deep sedation, analgesia and immobilization during surgery, as well as enhance post-operative recovery. Reduced muscle relaxant use during surgery poses the risk of inadequate immobilization during the operation, which may result in serious surgical complications. Intravenous bolus administration of fentanyl is currently the most popular method to maintain the depth of anesthesia during such operations. However, the side effects include intraoperative hypotension, bradycardia, and postoperative nausea and vomiting. The ultra-short acting remifentanil may be appropriate for inhibiting the bucking reflex during surgery, but the risk of opioid-induced hyperalgesia and opioid tolerance after surgery has been reported. In recent studies, intravenous lidocaine has been shown to increase the depth of anesthesia and provide analgesia, with no muscle relaxing effect.

The aim of this study is to examine the depth of anesthesia, surgical operating conditions, and the recovery profile with the use of a continuous lidocaine infusion.

DETAILED DESCRIPTION:
1. Purpose of the Study:

   This study is a single-center clinical trial in Taiwan, targeting the enrollment of 150 participants. The primary goal is to evaluate the effects of lidocaine infusion in thyroid surgery and to analyze whether it differs from or offers advantages over conventional anesthetic methods. As with any treatment, risks are involved, and clinical trials are no exception. Please carefully consider your participation in this trial.
2. Current Status of the Investigational Products:

   * Lidocaine (Local Anesthetic):

   Lidocaine is a commonly used local anesthetic for injection, as well as a routine intravenous anesthetic induction drug in general anesthesia. It is also frequently used to treat arrhythmias. Large-scale data analyses confirm its high safety profile. Continuous infusion has been shown to enhance intraoperative sedation and postoperative pain relief.

   -Fentanyl and Remifentanil (Systemic Analgesics): Fentanyl and its ultra-short-acting variant, remifentanil, are the most commonly used opioid analgesics in surgical anesthesia.
3. Inclusion and Exclusion Criteria:

   Physicians or research staff at our hospital will discuss the necessary conditions for participation with you. Please provide honest information about your medical history.
   * Inclusion Criteria:

   Age: 20-75 years Diagnosed with thyroid nodules or tumors Recommended for surgical excision by general surgeons or otolaryngologists Use of recurrent laryngeal nerve monitoring during surgery
   * Exclusion Criteria:

   High anesthesia risk Liver or kidney function impairment Known allergies to anesthetic drugs used in the surgery (Sevoflurane, Propofol, Lidocaine, Remifentanil, Fentanyl)
4. Study Methods and Procedures:

   -Preoperative Assessment: If you decide to join and sign the consent form, a routine preoperative health examination will be conducted, including blood and urine tests, height and weight measurements, heart rate and blood pressure monitoring, ECG, and chest X-rays.

   -Study Design:

   Participants will be randomly divided into three groups of 50 individuals. All participants will receive general anesthesia and intraoperative recurrent laryngeal nerve monitoring. Each group will have a different anesthesia and pain management approach:
   * Group P (Intermittent Fentanyl Infusion): Maintained with volatile anesthetic gas (sevoflurane) and intermittent fentanyl infusion.
   * Group L (Continuous Lidocaine Infusion): Maintained with sevoflurane and continuous lidocaine infusion.
   * Group R (Continuous Remifentanil Infusion): Maintained with sevoflurane and continuous remifentanil infusion.

   All other anesthesia procedures will follow routine clinical practice.

   During the surgery, the following will be monitored and recorded:

   -Intraoperative vital signs (heart rate, blood pressure, oxygen saturation)

   -Anesthesia parameters (e.g., inhaled anesthetic concentration, bispectral index(BIS) monitoring, neuromuscular response)

   -Surgery quality, occurrences of bucking, and duration Dosages of fentanyl, remifentanil, and lidocaine used

   Postoperative evaluations include:

   -Surgical environment quality assessed by the surgeon

   -Recovery scores using the Aldrete scoring system

   -Pain scores (VAS, 1-10) in the recovery room
   * Analgesic use within 24 hours post-surgery
   * On the first postoperative day, a nurse will assess recovery, side effects (e.g., sore throat, nausea), and pain levels. Appropriate treatments will be provided if necessary.
5. Potential Side Effects and Management:

   Risks Associated with Investigational Products:
   * Common (<10%):

   Circulatory: Mild bradycardia, slight increase in blood pressure Central nervous system(CNS): Paresthesia, dizziness Gastrointestinal: Mild nausea or vomiting -Uncommon (<1%): Central nervous system(CNS): Central nervous toxicity (seizures, perioral numbness, tongue numbness, auditory hypersensitivity, confusion, mild headache, tinnitus, slurred speech) -Rare (<0.1%): Severe allergic reactions: Anaphylactic shock Central nervous system(CNS): Neuropathy, peripheral nerve damage, arachnoiditis, unconsciousness, tremors Cardiac: Cardiac arrest, arrhythmias Respiratory: Respiratory depression
   * Management of Serious Adverse Effects:

   Immediately stop the local anesthetic infusion and provide emergency treatment for systemic toxicity symptoms.

   For seizures, administer anticonvulsants (e.g., thiopental 100-500 mg IV, diazepam 5-10 mg IV). If needed, administer suxamethonium for muscle relaxation.

   For cardiovascular instability, administer ephedrine (5-10 mg IV), and repeat if necessary.

   If cardiac arrest occurs, initiate cardiopulmonary resuscitation.
   * Risks of Routine General Anesthesia:

   Propofol (IV anesthetic): May cause mild bradycardia; very rarely (<0.0014%) may result in severe bradycardia.

   Sevoflurane (inhaled anesthetic): May cause mild bradycardia, hypotension, or postoperative nausea/vomiting (30-40%).

   Fentanyl/Remifentanil: May cause mild bradycardia, hypotension, or postoperative nausea/vomiting (10-50%).

   -Management: For severe bradycardia or hypotension, appropriate medications will be administered.

   For nausea or vomiting, antiemetics will be provided as needed.

   -If any severe side effects occur, please: Contact the 24-hour emergency hotline. Seek medical attention at the nearest emergency room if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-75 years old
* Receiving open thyroid surgery
* Using intraoperative neurophysiological monitoring

Exclusion Criteria:

* Allergic to opioids or lidocaine.
* Unsuitable for prolonged lidocaine infusion due to impaired cardiac function or severe arrhythmias.
* Impaired renal function (eGFR < 30).
* Liver dysfunction (Child-Pugh score B/C).

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
bucking and inadequate depth of anesthesia incidence | Perioperative
  participants bucking and inadequate depth of anesthesia incidence counts during the surgery

SECONDARY OUTCOMES:
Surgeon satisfaction | Perioperative
  Surgeon satisfaction during surgery in scale of 1-3, 1 as most-satisfied, 3 as unsatisfied.
Perioperative fentanyl usage | Perioperative
  Perioperative fentanyl usage
Post operative analgesia requirement | 24 hours postoperative
  Analgesia requirement during firs 24 hours after surgery
Perioperative hemodynamic stability | perioperative
  Perioperative hemodynamic stability(SBP with 20% compared to preoperative)
Prolonged sedation | Post operative to leaving PACU
  Record patient's consciousness level using Aldrete score: right after extubation, upon arrival at post anesthesia care unit(PACU)(10 minutes after surgery), and on leaving PACU(60 minutes after surgery).
VAS score while in post anesthesia care unit(PACU) | Post operative to leaving PACU
  VAS score while in PACU in 15 minutes, 30 minutes and 60 minues.
postoperative side effects (sore throat, postoperative nausea and vomiting etc.) | 24 hours postoperative
  postoperative side effects (sore throat, postoperative nausea and vomiting, etc.)

OTHER OUTCOMES:
dosage of fentanyl, remifentanil and lidocaine. | Perioperative
  dosage of fentanyl, remifentanil and lidocaine.

CONTACTS AND LOCATIONS:
Overall Officials: Zhen Xiu Chen, M.D., Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung veterans general hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 1 year after publication and ending 3 years after the publication of results
Access Criteria: describes planned analyses must be submitted

REFERENCES:
- [Background] Choi GJ, Kang H, Ahn EJ, Oh JI, Baek CW, Jung YH, Kim JY. Clinical Efficacy of Intravenous Lidocaine for Thyroidectomy: A Prospective, Randomized, Double-Blind, Placebo-Controlled Trial. World J Surg. 2016 Dec;40(12):2941-2947. doi: 10.1007/s00268-016-3619-6. PMID 27379388
- [Background] De Oliveira GS Jr, Fitzgerald P, Streicher LF, Marcus RJ, McCarthy RJ. Systemic lidocaine to improve postoperative quality of recovery after ambulatory laparoscopic surgery. Anesth Analg. 2012 Aug;115(2):262-7. doi: 10.1213/ANE.0b013e318257a380. Epub 2012 May 14. PMID 22584558
- [Background] De Oliveira GS Jr, Duncan K, Fitzgerald P, Nader A, Gould RW, McCarthy RJ. Systemic lidocaine to improve quality of recovery after laparoscopic bariatric surgery: a randomized double-blinded placebo-controlled trial. Obes Surg. 2014 Feb;24(2):212-8. doi: 10.1007/s11695-013-1077-x. PMID 24036842
- [Background] Beaussier M, Delbos A, Maurice-Szamburski A, Ecoffey C, Mercadal L. Perioperative Use of Intravenous Lidocaine. Drugs. 2018 Aug;78(12):1229-1246. doi: 10.1007/s40265-018-0955-x. PMID 30117019
- [Background] Lee JH, Koo BN, Jeong JJ, Kim HS, Lee JR. Differential effects of lidocaine and remifentanil on response to the tracheal tube during emergence from general anaesthesia. Br J Anaesth. 2011 Mar;106(3):410-5. doi: 10.1093/bja/aeq396. Epub 2011 Jan 2. PMID 21205628
- [Background] Fletcher D, Martinez V. Opioid-induced hyperalgesia in patients after surgery: a systematic review and a meta-analysis. Br J Anaesth. 2014 Jun;112(6):991-1004. doi: 10.1093/bja/aeu137. PMID 24829420
- [Background] Hsieh CY, Tan H, Huang HF, Huang TY, Wu CW, Chang PY, Lu DV, Lu IC. Optimization of Intraoperative Neural Monitoring of the Recurrent Laryngeal Nerve in Thyroid Surgery. Medicina (Kaunas). 2022 Mar 30;58(4):495. doi: 10.3390/medicina58040495. PMID 35454334
- [Background] Govindarajan R, Shah A, Ravikumar S, Reddy SK, Kannan U, Mukerji AN, Cherian JG, Foster C, Livingstone D. Lidocaine Infusion Improves the Functionality of Intraoperative Nerve Monitoring During Thyroid Surgery: A Prospective, Randomized, Double-Blinded Study. J Clin Med Res. 2021 Apr;13(4):214-221. doi: 10.14740/jocmr4458. Epub 2021 Apr 27. PMID 34007359